CLINICAL TRIAL: NCT02844179
Title: (+)-Alpha-Dihydrotetrabenazine Phase I
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kirk A. Frey (Other)
Collaborators: Adeptio Pharmaceuticals (Unknown)
Responsible Party: Sponsor-Investigator, Kirk A. Frey, Professor of Radiology, University of Michigan
Organization: University of Michigan (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00105810 -1
Record Dates: First submitted 2016-07-20; First posted 2016-07-26 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- dose escalation (Experimental): Single dose administration of (+)-alpha-Dihydrotetrabenazine (HTBZ), escalating dosage amounts 7.5 - 30 mg orally
  Interventions: Drug: HTBZ

INTERVENTIONS:
Drug: HTBZ

SUMMARY:
This research study is intended to determine the initial safety and tolerability of single oral doses of the drug (+)-alpha-dihydrotetrabenaxine (HTBZ) in normal volunteers. HTBZ is believed to be the active ingredient in the FDA-approved drug tetrabenazine (TBZ, brand name Xenazine), prescribed for treatment of involuntary movements in patients with Huntington's chorea. TBZ is a mixture of closely-related compounds (isomers) and is readily metabolized (converted) in the human body to HTBZ and related isomers. Investigators believe that HTBZ, the drug to be studied in this research, is the active ingredient in TBZ. The present study will confirm safety and tolerability of HTBZ and will investigate its expected effects on brain sites that are the target of TBZ therapy.

ELIGIBILITY:
Inclusion Criteria:

* able to provide informed consent

Exclusion Criteria:

* pregnant or lactating female subjects
* Subjects taking medications that interfere with VMAT2 (ex amphetamine)
* History of significant neurologic or psychiatric conditions
* Significant active medical conditions
* Alcohol or illicit substance use or dependence

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-07; Primary Completion 2017-06-27 (Actual); Study Completion 2017-06-27 (Actual)

PRIMARY OUTCOMES:
VMAT2 occupancy by HTBZ determined by positron emission tomography (PET) scanning | 60 minutes post-administration of HTBZ

CONTACTS AND LOCATIONS:
Overall Officials: Kirk A Frey, MD, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan hospitals, Ann Arbor, Michigan, United States